CLINICAL TRIAL: NCT01413568
Title: A Phase I/II Study Evaluating the Safety and Efficacy of Intravenous POL6326 for the Mobilization and Transplantation of HLA-Matched Sibling Donor Hematopoietic Stem Cells in Patients With Advanced Hematological Malignancies
Brief Title: Safety and Efficacy of POL6326 for Mobilization/Transplant of Sibling Donor in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201112026; POL-4 (Other: Polyphor)
Record Dates: First submitted 2011-08-05; First posted 2011-08-10 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myeloid Leukemia in Remission; Adult Acute Lymphoblastic Leukemia in Remission; Chronic Myelogenous Leukemia (CML); Non-Hodgkin's Lymphoma (NHL) or Hodgkin's Disease (HD) in 2nd or Greater Complete Remission, Partial Remission; Chronic Lymphocytic Leukemia (CLL); Multiple Myeloma (MM); Myelodysplastic Syndrome (MDS); Myeloproliferative Disorders
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — balixafortide; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donor (Phase I and Phase II) (Experimental): On Day 1 (and possibly Day 2) POL6326 IV Infusion with increasing dose levels in Phase I or with random dose assignment (from the 2 selected from Phase I) in phase II
  Leukapheresis collection on Day 1 (and possibly Day 2)
  Interventions: Drug: POL6326; Procedure: Leukapheresis
- Recipient (Experimental): Day 0 - PBSC transplant with stem cells mobilized with IV POL6326
  Interventions: Procedure: PBSC Transplant

INTERVENTIONS:
Drug: POL6326
  Arms: Donor (Phase I and Phase II)
Procedure: Leukapheresis
  Arms: Donor (Phase I and Phase II)
Procedure: PBSC Transplant
  Arms: Recipient

SUMMARY:
Determine the safety and tolerability of POL6326 when used as a single mobilization agent.

DETAILED DESCRIPTION:
Current protocols use G-CSF to mobilize hematopoietic progenitor cells from matched sibling donors. This process requires from four to six days of G-CSF injection and is associated with significant morbidity, most notably bone pain. POL6326 is associated with few side effects and collection of cells occurs on the same day as POL6326 administration.

This study will evaluate the safety and efficacy of this novel agent for hematopoietic progenitor cell mobilization and allogeneic transplantation based on the following hypotheses:

1. Donors mobilized with intravenous POL6326 will require fewer collections than have previously been seen for donors mobilized with subcutaneous plerixafor.
2. Healthy HLA-matched donors receiving one or two infusions of POL6326 will mobilize sufficient CD34+ cells (at least 2.0 x 106 CD34+ cells/kg recipient weights) following leukapheresis to support a hematopoietic cell transplant.
3. IV POL6326 will result in more rapid kinetics and a higher maximum (peak) of human CD34+ stem cells mobilized from human normal allogeneic donors compared to previous donors who were mobilized with plerixafor.
4. The hematopoietic cells mobilized by IV POL6326 will be functional and will result in prompt and durable hematopoietic engraftment following transplantation into HLA-identical siblings with advanced hematological malignancies using various non-myeloablative and myeloablative conditioning regimens and regimens for routine GVHD prophylaxis.

ELIGIBILITY:
Donor Inclusion Criteria

* Donor must be 18 to 70 years of age inclusive.
* Donor must be a 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* Donor must have adequate cardiac function with no history of congestive heart failure and no history of atrial fibrillation or ventricular tachyarrhythmia.
* Donor must have adequate renal function as defined by a minimum creatinine clearance (CrCl) value of >30 ml/min.
* Donor must have adequate hepatic function as defined by a total bilirubin <3x upper limit of normal.
* Donor must have adequate neurologic function as defined by NO evidence of a severe central or peripheral neurologic abnormality and no history of cerebrovascular accident or seizure disorder requiring anticonvulsant medication.
* Donor must be HIV-1&2 antibody and HTLV-1&2 antibody sero-negative by FDA licensed test.
* Donor must have an ECOG performance status of 0 or 1.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Donor must demonstrate ability to be compliant with study regimen.
* Donor must be able to understand and willing to sign an IRB approved written informed consent document.

Recipient Inclusion Criteria

* Recipient must have available the successful collection of a POL62326 mobilized product.
* Recipient must be 18 to 75 years of age inclusive.
* Recipient must have a 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Recipient must have one of the following diagnoses:
* Acute myelogenous leukemia (AML) in 1st or subsequent remission
* Acute lymphoblastic leukemia (ALL) in 1st or subsequent remission
* Chronic myelogenous leukemia (CML)
* Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete remission, partial remission
* Chronic lymphocytic leukemia (CLL)
* Multiple myeloma (MM)
* Myelodysplastic syndrome (MDS)
* Myeloproliferative disorder (MPD)
* Recipient must have adequate cardiac function with a left ventricular ejection fraction > 40%.
* Recipient must have adequate pulmonary function defined as NO severe or symptomatic restrictive or obstructive lung disease, and formal pulmonary function testing showing an FEV1 >50% (predicted) and a DLCO >40% (predicted), corrected for hemoglobin.
* Recipient must have adequate hepatic function as defined by a total bilirubin <3x upper limit of normal or absence of hepatic fibrosis/cirrhosis.
* Recipient must have adequate neurologic function as defined by NO evidence of a severe central or peripheral neurologic abnormality. Patients with a history of previous CNS tumor involvement are eligible provided they are without symptoms or signs and the CNS is now free of disease on lumbar puncture and CT scan of the brain.
* Recipient must be HIV-1&2 antibody and HTLV-1&2 antibody sero-negative by FDA licensed test.
* Recipient must have an ECOG performance status of 0 or 1.
* Recipient must demonstrate ability to be compliant with medical regimen.
* Recipient must have life expectancy of greater than 2 months.
* Recipient must be able to understand and willing to sign an IRB approved written informed consent document.

Donor Exclusion Criteria

* Donor must not have an active infection at the time of study entry.
* Donor must not have active alcohol or substance abuse within 6 months of study entry.
* Donor must not be currently enrolled on another investigational agent study.
* Donor must not have any medical condition, which, in the opinion of the clinical investigator, would interfere with his/her evaluation.
* Donor must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* If female and of child-bearing age, donor must not be pregnant or breastfeeding.

Recipient Exclusion Criteria

* Recipient must not have had (the following therapies within the following timeframe):
* Investigative drugs within 21 days
* Recipient must have no evidence of active infection at the time of the transplant preparative regimen or at time of transplantation.
* Recipient must have no active alcohol or substance abuse within 6 months of study entry.
* Recipient must not be pregnant and/or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Phase I Study - safety and tolerability of POL6326 as a mobilization agent. | 30 days
Phase II Study - determine the number of allogeneic donors who require a second leukapheresis | 2 days
  Determine the number of allogeneic donors which collect >= 2 mill CD34+ cells with one or two leukapheresis procedures treated with IV POL6326. Comparison with historic group of donors who were mobilized with 240 µg/kg SC plerixafor.

SECONDARY OUTCOMES:
Phase I Study - define maximum tolerated dose of POL6326 | 30 days
Phase II Study - the proportion of HLA-identical sibling donors who experience grade 3-4 infusional toxicity and the proportion who are safely mobilized | 30 days
  To estimate the proportion of HLA-identical sibling donors who experience grade 3-4 infusional toxicity and the proportion from whom > 2 mill CD34+ cells/kg recipient weight are safely mobilized following one or two leukapheresis procedures
Phase II Study - pharmacokinetics and pharmacodynamics of IV POL6326 | Day 1-3
  Stem cell and T-cell phenotyping
Phase II Study - rate of acute GVHD and chronic GVHD in patients who receive IV POL6326 mobilized peripheral blood stem cells. | Day 100 (+/- 7 days) or Day 365 (+/-14 days)
  Acute GVHD - Day 100 (+/- 7 days) Chronic GVHD - Day 365 (+/- 14 days)
Phase II Study - kinetics of neutrophil and platelet engraftment in recipients of POL6326 mobilized peripheral blood stem cells. | Day 365 (+/- 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Couriel, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Washington University School of Medicine, St Louis, Missouri